CLINICAL TRIAL: NCT06089122
Title: Efficacy, Safety, and Pharmacokinetics of Shu Yang IVIG in Patients With Primary Immunodeficiency
Brief Title: Efficacy, Safety, and Pharmacokinetics of Shu Yang IVIG
Acronym: Imunoforte
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Collaborators: Sichuan Yuanda Shuyang Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMUNOFORTE; U1111-1298-7059 (Other: WHO)
Record Dates: First submitted 2023-09-19; First posted 2023-10-18 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-10

CONDITIONS: Primary Immunodeficiency Disease
Keywords: IVIG; IMUNOFORTE; PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: Patients with primary immunodeficiency will switch to Shu Yang IVIG and optimize the posology in a run-in period of 2 to 6 administrations. In the one-year test period, the patients will receive the test IVIG at 21- or 28-day intervals and be followed. IgG trough levels will be collected at all visits. At Visit 4, at least 20 patients will perform the PK assessment, collecting additional blood samples.
Masking Description: The trial will be open-label and single-arm. Therefore, there will be no randomization or blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IVIG (Experimental): Patients with primary immunodeficiency will switch to Shu Yang IVIG and optimize the posology to IgG 300 to 600 mg every 21 or 28 days in a run-in period of 2 to 6 administrations, aiming at keeping the IgG trough levels above 5 g/L. In the one-year test period, the patients will receive the test IVIG at the same dose/intervals of the optimization. However, the IgG trough levels will be monitored every visit, and new adjustments/dose optimization will be performed whenever needed to keep the IgG trough levels above 5g/L.
  Interventions: Biological: IVIG

INTERVENTIONS:
Biological: IVIG — Patients with primary immunodeficiency will switch to Shu Yang IVIG and optimize the posology to IgG 300 to 600 mg every 21 or 28 days in a run-in period of 2 to 6 administrations, aiming at keeping the IgG trough levels above 5 g/L. At Visit 4, at least 20 patients will perform the PK assessment, collecting additional blood samples.
  Other Names: Shu Yang IVIG

SUMMARY:
To evaluate the safety, efficacy, and pharmacokinetic properties of Shu Yang intravenous immune globulin in patients with primary immune deficiency aged less than 60 years.

The main benefit of IVIG is to help the body fight against a large variety of infections generally associated with morbidity and mortality in patients with primary immunodeficiency diseases, particularly in CVID and XLA. In addition, a decrease in the number of infections, a reduction in medications and hospitalizations, and a better quality of life are expected.

Throughout treatment, approximately one-fourth of persons may experience a side effect. These are usually mild or bothersome but not dangerous. Very rarely, more serious side effects like allergic reactions or low blood counts (anemia) can occur. One of the most common side effects is headache. Other side effects include chills, fever, flushing, flu-like muscle pains or joint pains, feeling tired, nausea, vomiting, and rash. For the most part, these reactions typically happen with the first dose of IVIG or because change to a different brand of IVIG. All IVIG products have similar warnings and contraindications, such as the potential for renal failure, thrombotic events, aseptic meningitis, hemolysis, and anaphylactic reactions.

DETAILED DESCRIPTION:
This is a Phase III, open-label, prospective, single-arm, multicenter trial to evaluate the efficacy of IVIG in maintaining the average of severe bacterial infections in less than one per year. The safety and pharmacokinetics (PK) of the investigational product will also be evaluated. Fifty male or female patients aged up to 60 years old will be selected. At least 20 patients must be up to 17 years old. During the trial, at least 20 adult patients will be invited to make up the PK assessment subgroups.

After obtaining the signed Informed Consent/Assent Form , the screening procedures will be performed including the immune deficiency history from the medical records and safety exams. Patients will start the trial with a run-in period to stabilize the IgG trough levels. This period could last two to six visits with posological adjustments until the last two IgG trough levels are above 4 (5) g/L.

After the run-in, the one-year test period will start at the V0. Depending on the treatment regimen, the patients will receive IVIG every 21 days (±3 days) up to day 378 or every 28 days (±4 days) up to day 364 when the close-out visit will occur. In all visits from all patients, a blood sample will be collected immediately before each IVIG administration to assess the IgG trough levels.

To assess the investigational product PK properties, a group of 20 patients will collect additional blood samples for dosing IgG levels between Visit 4 and Visit 5. Those taking IVIG every 21 days, will collect six additional blood samples at the following times after the injection 30 min, 2h, 24h, 72h, 7 days, and 14 days. Those taking IVIG every 28 days will collect seven additional blood samples at the times 30 min, 2h, 24h, 72h, 7 days, 14 days, and 21 days.

Adverse events will be collected at all visits to fulfill the safety endpoints. Moreover, the patients will have continuous access to the investigator's team to report adverse events, be instructed about how to proceed, or even perform Extra visits for presential medical evaluation.

Additionally, the patient will receive a diary to record AEs, any medication taken, infections of any kind, days of hospitalization, and days missed from major activities due to infections.

Trial duration: Each patient can participate in the trial for a maximum period of approximately 540 days from the time of signing the ICF or IAF until the close-out visit, including a Run-in period, depending on treatment regimen.

Blinding and Randomization: This is an open-label trial; no blinding and randomization procedures will be applied.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent.
2. Male or female.
3. Ages ≤ 60 years old and ≥ 06 years old.
4. Diagnosis of Primary Immunodeficiency Disease (PID) with a reduction in antibody production due to:

   a. Common Variable Immunodeficiency (CVID) as per European Immunodeficiency Society (ESID)/Pan American Immunodeficiency Group (PAGID), as defined in section 5.1, OR b. X-linked agammaglobulinemia (XLA) as per ESID/PAGID, as defined in section 5.1.
5. Receiving replacement therapy with intravenous immunoglobulin at 21- to 28-day intervals at 300-600 mg/kg/month for a minimum of 2 months before the start of the study;
6. Absence of episodes of serious bacterial infections with previous use of an IV immunoglobulin for at least 3 months before screening;
7. Negative pregnancy test (in female patients with childbearing potential); readiness to use reliable methods of contraception throughout the study period;
8. Patients who participated in a clinical trial with another experimental IVIG may be enrolled if they have a potential benefit according to Res. CNS 251/1997;
9. Patients currently on treatment with any subcutaneous or intramuscular immunoglobulin may be enrolled switching to IVIG therapy at the investigator's discretion, considering the potential benefit to the patient.

Exclusion Criteria:

1. Known intolerance or hypersensitivity to immunoglobulins or components of the test article;
2. Any contraindications to the use of immunoglobulins;
3. Secondary immunodeficiency or conditions potentially causing secondary immunodeficiency such as chronic lymphoid leukemia, lymphoma, multiple myeloma, protein-losing enteropathies or nephropathies, and hypoalbuminemia;
4. Clinically relevant changes in the safety exams are defined as:

   * Blood count

     o Hb < 10.5 g/dL

     o Leukocytes < 3,000 /uL or >10,000 cells / uL

     o Absolute neutrophil count < 1,000 cells/mm3;
   * Coagulation o TP and aPTT > 2.5 x ULN
   * Biochemistry o glycated hemoglobin > 6.5%

     * total bilirubin and fractions, alkaline phosphatase, ALT, AST, GGT > 2.5 x ULN
     * creatinine above 3mg/dl or creatinine clearance < 30mL/min
   * Urine I.

     * Leukocyturia > 10,000 cells/mL 5. Any cancer either active or resolved within the last 12 months before screening;

6. Receiving any blood products (except intravenous immunoglobulins) during the last 3 months before screening;

7. Any febrile illness within 14 days before enrollment; Note: The patient may be rescreened after recovery.

8. History of thrombotic events (including myocardial infarction, stroke, pulmonary embolism, and deep vein thrombosis) within 6 months before enrollment;

9. Previous use of live attenuated virus vaccines;

10. Selective deficiency of immunoglobulin A (IgA) or known antibodies to IgA;

11. Known drug or alcohol abuse;

12. The need to use other investigational drugs, systemic immunosuppressants, and any other immunoglobulins;

13. Pregnancy or lactation;

14. Inability to comply with the protocol activities;

15. PIDs other than CVID or X-linked agammaglobulinemia

16. Patients infected with HIV, HBV or HCV

17. Patients with AIDS, cystic fibrosis, or active hepatitis B or C.

18. Any other condition that, in the Investigator's opinion may increase the risk of participation in this study.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-01-08 (Estimated); Study Completion 2025-06-08 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Objective (average of acute serious bacterial infections) | Between Visit 0 and Final Visit (through study completion, an average of 1 year)
  The incidence of serious bacterial infections (septicemia, meningitis, visceral abscess, osteomyelitis, and pneumonia) within the 1-year follow-up is less than 1.0 per patient/year in the average of the population.

SECONDARY OUTCOMES:
Secondary Efficacy Objectives (assessment of the rate of non-serious infections) | Average incidence of non-serious infections per patient between Visit 0 and Final Visit (through study completion, an average of 1 year), as documented as treatment emergent adverse events (TEAEs);
  The incidence of all acute infections except the serious acute bacterial infections within the 1-year follow-up (simple descriptive statistics).
Secondary Efficacy Objectives | Average number of days for treating infections per patient between visit 0 and final visit (through study completion, an average of 1 year), as documented as treatment emergent adverse events (TEAEs);
  Assessment of treatment length of infections per year;
Secondary Efficacy Objectives | Average number of days off from school/work per patient/month, as documented in the patient's diary (through study completion, an average of 1 year);
  Assessment of missing time from school/work due to infections per month;
Secondary Efficacy Objectives | Number of days hospitalized per month overall and due to infection, as documented as treatment emergent adverse events - TEAEs (through study completion, an average of 1 year).
  Assessment of hospitalization episodes and length.

OTHER OUTCOMES:
Secondary Pharmacokinetic (PK) Objectives | 9 months
  To assess the total IgG serum concentration before each infusion (IgG trough levels), between Visit 4 and Final Visit (through study completion).
Secondary Pharmacokinetic (PK) Objectives | 28 days
  To assess total serum IgG profile (concentration vs time) at specific times between the 5th and 6th infusion
IgG half-life | 28 days
  Determine IgG half-life from concentration vs time curve
Area under the IgG curve | 28 days
  Determine IgG AUC from concentration vs time curve
IgG distribution volume | 28 days
  Determine IgG Vd from concentration vs time curve
IgG elimination constant | 28 days
  Determine IgG Kel from concentration vs time curve
Incidence, severity, and causality of adverse events | 1, 24, and 72 hours after each infusion (through study completion, an average of 1 year);
  Assessment of infusion-related adverse events;
Secondary Safety Objective | Incidence, severity, and causality of all treatment-emergent adverse events, except those infusion-related (through study completion, an average of 1 year).
  Assessment of treatment emergent adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Ferrara, Study Director — Azidus Brasil

IPD SHARING:
Plan to Share IPD: No
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data of the study will become public

REFERENCES:
- [Background] Bierry G, Boileau J, Barnig C, Gasser B, Korganow AS, Buy X, Jeung MY, Roy C, Gangi A. Thoracic manifestations of primary humoral immunodeficiency: a comprehensive review. Radiographics. 2009 Nov;29(7):1909-20. doi: 10.1148/rg.297095717. PMID 19926753
- [Background] Blasczyk R, Westhoff U, Grosse-Wilde H. Soluble CD4, CD8, and HLA molecules in commercial immunoglobulin preparations. Lancet. 1993 Mar 27;341(8848):789-90. doi: 10.1016/0140-6736(93)90563-v. PMID 8096001
- [Background] Bonilla FA, Barlan I, Chapel H, Costa-Carvalho BT, Cunningham-Rundles C, de la Morena MT, Espinosa-Rosales FJ, Hammarstrom L, Nonoyama S, Quinti I, Routes JM, Tang ML, Warnatz K. International Consensus Document (ICON): Common Variable Immunodeficiency Disorders. J Allergy Clin Immunol Pract. 2016 Jan-Feb;4(1):38-59. doi: 10.1016/j.jaip.2015.07.025. Epub 2015 Nov 7. PMID 26563668
- [Background] BRUTON OC. Agammaglobulinemia. Pediatrics. 1952 Jun;9(6):722-8. No abstract available. PMID 14929630
- [Background] Busse PJ, Razvi S, Cunningham-Rundles C. Efficacy of intravenous immunoglobulin in the prevention of pneumonia in patients with common variable immunodeficiency. J Allergy Clin Immunol. 2002 Jun;109(6):1001-4. doi: 10.1067/mai.2002.124999. PMID 12063531
- [Background] Cordero E, Goycochea-Valdivia W, Mendez-Echevarria A, Allende LM, Alsina L, Bravo Garcia-Morato M, Gil-Herrera J, Gudiol C, Len-Abad O, Lopez-Medrano F, Moreno-Perez D, Munoz P, Olbrich P, Sanchez-Ramon S, Soler-Palacin P, Aguilera Cros C, Arostegui JI, Badell Serra I, Carbone J, Fortun J, Gonzalez-Granado LI, Lopez-Granados E, Lucena JM, Parody R, Ramakers J, Regueiro JR, Riviere JG, Roca-Oporto C, Rodriguez Pena R, Santos-Perez JL, Rodriguez-Gallego C, Neth O. Executive Summary of the Consensus Document on the Diagnosis and Management of Patients with Primary Immunodeficiencies. J Allergy Clin Immunol Pract. 2020 Nov-Dec;8(10):3342-3347. doi: 10.1016/j.jaip.2020.05.008. PMID 33161963
- [Background] Hagan JB, Fasano MB, Spector S, Wasserman RL, Melamed I, Rojavin MA, Zenker O, Orange JS. Efficacy and safety of a new 20% immunoglobulin preparation for subcutaneous administration, IgPro20, in patients with primary immunodeficiency. J Clin Immunol. 2010 Sep;30(5):734-45. doi: 10.1007/s10875-010-9423-4. Epub 2010 May 8. PMID 20454851
- [Background] Hartung HP, Mouthon L, Ahmed R, Jordan S, Laupland KB, Jolles S. Clinical applications of intravenous immunoglobulins (IVIg)--beyond immunodeficiencies and neurology. Clin Exp Immunol. 2009 Dec;158 Suppl 1(Suppl 1):23-33. doi: 10.1111/j.1365-2249.2009.04024.x. PMID 19883421
- [Background] Herriot R, Sewell WA. Antibody deficiency. J Clin Pathol. 2008 Sep;61(9):994-1000. doi: 10.1136/jcp.2007.051177. PMID 18755724
- [Background] Hoffmann F, Grimbacher B, Thiel J, Peter HH, Belohradsky BH; Vivaglobin Study Group. Home-based subcutaneous immunoglobulin G replacement therapy under real-life conditions in children and adults with antibody deficiency. Eur J Med Res. 2010 Jun 28;15(6):238-45. doi: 10.1186/2047-783x-15-6-238. PMID 20696632
- [Background] IDF Guide for Nurses - Immunoglobulin Therapy for Primary Immunodeficiency Diseases. 4th, pp. 59.
- [Background] Milito C, Pulvirenti F, Pesce AM, Digiulio MA, Pandolfi F, Visentini M, Quinti I. Adequate patient's outcome achieved with short immunoglobulin replacement intervals in severe antibody deficiencies. J Clin Immunol. 2014 Oct;34(7):813-9. doi: 10.1007/s10875-014-0081-9. Epub 2014 Jul 22. PMID 25047154
- [Background] Mouthon L, Kaveri SV, Spalter SH, Lacroix-Desmazes S, Lefranc C, Desai R, Kazatchkine MD. Mechanisms of action of intravenous immune globulin in immune-mediated diseases. Clin Exp Immunol. 1996 May;104 Suppl 1:3-9. PMID 8625540
- [Background] Orange JS, Hossny EM, Weiler CR, Ballow M, Berger M, Bonilla FA, Buckley R, Chinen J, El-Gamal Y, Mazer BD, Nelson RP Jr, Patel DD, Secord E, Sorensen RU, Wasserman RL, Cunningham-Rundles C; Primary Immunodeficiency Committee of the American Academy of Allergy, Asthma and Immunology. Use of intravenous immunoglobulin in human disease: a review of evidence by members of the Primary Immunodeficiency Committee of the American Academy of Allergy, Asthma and Immunology. J Allergy Clin Immunol. 2006 Apr;117(4 Suppl):S525-53. doi: 10.1016/j.jaci.2006.01.015. PMID 16580469
- [Background] Pourpak Z, Aghamohammadi A, Sedighipour L, Farhoudi A, Movahedi M, Gharagozlou M, Chavoshzadeh Z, Jadid L, Rezaei N, Moin M. Effect of regular intravenous immunoglobulin therapy on prevention of pneumonia in patients with common variable immunodeficiency. J Microbiol Immunol Infect. 2006 Apr;39(2):114-20. PMID 16604243
- [Background] Primary immunodeficiency diseases. Report of an IUIS Scientific Committee. International Union of Immunological Societies. Clin Exp Immunol. 1999 Oct;118 Suppl 1(Suppl 1):1-28. doi: 10.1046/j.1365-2249.1999.00109.x. No abstract available. PMID 10540200
- [Background] Quinti I, Soresina A, Guerra A, Rondelli R, Spadaro G, Agostini C, Milito C, Trombetta AC, Visentini M, Martini H, Plebani A, Fiorilli M; IPINet Investigators. Effectiveness of immunoglobulin replacement therapy on clinical outcome in patients with primary antibody deficiencies: results from a multicenter prospective cohort study. J Clin Immunol. 2011 Jun;31(3):315-22. doi: 10.1007/s10875-011-9511-0. Epub 2011 Mar 2. PMID 21365217
- [Background] Radosevich M, Burnouf T. Intravenous immunoglobulin G: trends in production methods, quality control and quality assurance. Vox Sang. 2010 Jan;98(1):12-28. doi: 10.1111/j.1423-0410.2009.01226.x. Epub 2009 Jul 29. PMID 19660029
- [Background] Salehzadeh M, Aghamohammadi A, Rezaei N. Evaluation of immunoglobulin levels and infection rate in patients with common variable immunodeficiency after immunoglobulin replacement therapy. J Microbiol Immunol Infect. 2010 Feb;43(1):11-7. doi: 10.1016/S1684-1182(10)60002-3. Epub 2010 Mar 29. PMID 20434118
- [Background] Suri D, Rawat A, Singh S. X-linked Agammaglobulinemia. Indian J Pediatr. 2016 Apr;83(4):331-7. doi: 10.1007/s12098-015-2024-8. Epub 2016 Feb 24. PMID 26909497
- [Background] WHO. WHO RECOMMENDATIONS FOR THE PRODUCTION, CONTROL AND REGULATION OF HUMAN PLASMA FOR FRACTIONATION. pp. 69.
- [Background] Yazdani R, Habibi S, Sharifi L, Azizi G, Abolhassani H, Olbrich P, Aghamohammadi A. Common Variable Immunodeficiency: Epidemiology, Pathogenesis, Clinical Manifestations, Diagnosis, Classification, and Management. J Investig Allergol Clin Immunol. 2020;30(1):14-34. doi: 10.18176/jiaci.0388. Epub 2019 Feb 11. PMID 30741636